CLINICAL TRIAL: NCT04542967
Title: Convalescent Plasma as a Treatment for Patients With Severe COVID-19 Disease
Brief Title: Study on the Safety and Efficacy of Convalescent Plasma in Patients With Severe COVID-19 Disease
Acronym: PC-COVID-HCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Central Militar (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 047/2020
Record Dates: First submitted 2020-09-04; First posted 2020-09-09 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-09

CONDITIONS: Severe COVID-19 Disease
Keywords: SARS-CoV2; Convalescent Plasma; Severe Acute Respiratory Syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Biological Products

STUDY DESIGN:
Intervention Model Description: The PC-COVID-HCM clinical trial is a randomized, controlled, single-blind study .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research was blinded as possible for the result's evaluators and those responsible for the statistical analysis. All patients admitted to the investigation were placed with a marker indicating that they were a patient of the plasma protocol, but not mention the study group. The data collectors and the outcome adjudicators were unaware of the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): They will receive the standard care for critically ill inpatients.
- Convalescent plasma group. (Experimental): They will receive standard care for patients with severe COVID-19 disease and convalescent plasma disease.
  Interventions: Biological: Biological

INTERVENTIONS:
Biological: Biological — An administration unit of 200 ml convalescent plasma intravenous infusion every 24 hours for two doses.
  If a third dose of convalescent plasma is necessary, it may be used, as long as an evaluation of the research team is carried out.
  Other Names: Convalescent plasma
  Arms: Convalescent plasma group.

SUMMARY:
Currently, there is no specific treatment or vaccine for SARS-CoV-2 available, some drugs are being investigated as treatment, but the effect is unknown. A strategy and other method used before, in coronavirus pandemic (SARS-CoV in 2003 and MERS-CoV in 2012), was the use of immune (convalescent) plasma. Passive administration of antibodies through convalescent plasma transfusion may offer the only short-term strategy available to confer immediate immunity and being a relative immediately resource available for treat COVID-19 disease. This research proposes the passive administration of antibodies through the transfusion of convalescent plasma, in patients with severe COVID-19 disease.

DETAILED DESCRIPTION:
A randomized clinical trial comparing administration convalescent plasma to standard therapy for severe COVID-19 disease. Patients will be randomized 1:1 in a single blind study. The patients with SARS-CoV-2 PCR confirmed infection with pulmonary infiltrates and hypoxemia will be screened and invited to participate. Our primary outcomes will be disease progression and mortality, evaluate of ordinal Scale for Clinical Improvement and. (WHO)

ELIGIBILITY:
Inclusion Criteria:

* O2 saturation <93%
* Radiographic evidence of moderate pneumonia according to Rale's classification.
* Acute respiratory distress syndrome (PaO2 / FiO2 <300 or SpO2 / FiO2 ≤ 315)
* Authorization to participate in the study and have informed consent letter, signed by the patient or the person responsible for the patient in case of critical patients (intubated)

Exclusion Criteria:

* Pregnant patients
* History of transfusion reactions
* Patients with congestive heart failure
* Patients with a history of chronic kidney failure on dialysis
* Patients with multiple organ failure
* Patients who does not accept or agree with the treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Disease progression | Up to 30 days later from study entry
  Change in ordinal Scale for Clinical Improvement (WHO). The progression disease, its the change in the severity score; a bigger number to the obtained after randomization
Side effects | Up to 30 days later from study entry
  Side effects associated with the administration of convalescent plasma
Mortality | Up to 30 days later from study entry
  Any cause of death

SECONDARY OUTCOMES:
Respiratory improvement | 10 days
  Change in partial pressure of arterial Oxygen to Fraction of inspired Oxygen ratio (PaO2/FiO2)
Clinical improvement | 10 days
  Change in oxygen saturation levels
Acute adverse events (AAE) | After receiving intervention, an average time one hour, until 24 hours after administration.
  Transfusion reactions during transfusion.

OTHER OUTCOMES:
Inflammatory biomarkers (D dimer) | 10 days
  Change in pro-inflammatory biomarkers (D dimer μg/l)
Inflammatory biomarkers (Ferritin) | 10 days
  Change in pro-inflammatory biomarkers ( Ferritin μg/L )
Inflammatory biomarkers (CPR) | 10 days
  Change in pro-inflammatory biomarkers, C-reactive protein ( CPR mg/L )
Inflammatory biomarkers (LDH) | 10 days
  Change in pro-inflammatory biomarkers, lactate dehydrogenase ( LDH UI/L)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen G Torres, MD, Principal Investigator — Hospital Central Militar
Locations (1):
- Hospital Central Militar, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Plan to make IPD still not decided and would need approval by regulatory authorities
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 6 months after publication
Access Criteria: PRIOR APPLICATION

REFERENCES:
- See also: Clinical Characteristics of Coronavirus Disease 2019 in China — http://pubmed.ncbi.nlm.nih.gov/32109013/
- See also: Potential interventions for novel coronavirus in China: A systematic review — http://pubmed.ncbi.nlm.nih.gov/32052466/
- See also: Use of convalescent plasma therapy in SARS patients in Hong Kong — http://pubmed.ncbi.nlm.nih.gov/15616839/